CLINICAL TRIAL: NCT03263780
Title: High-Resolution, 18F-fluciclovine PET-MRI for Mapping Prostate Cancer in Patients Considering Focal High-Intensity Focused Ultrasound (HIFU) Therapy
Brief Title: High Resolution PET-MRI Before Prostate Cancer HIFU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Timothy J. Daskivich (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor-Investigator, Timothy J. Daskivich, Staff Physician I, Division of Urology; Urologic Oncologist; Director, Health Services Research, Department of Surgery Cedars Sinai Medical Center, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IIT2016-19-DASKIVICH-18F
Record Dates: First submitted 2017-08-22; First posted 2017-08-28 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: Diagnostic imaging; High-Intensity Focused Ultrasound; HIFU; 18F-Fluciclovine; high resolution diffusion-weighted imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-Fluciclovine (Experimental): 10mCi +/-20% 18F-fluciclovine injection
  Interventions: Drug: 18F-Fluciclovine

INTERVENTIONS:
Drug: 18F-Fluciclovine — Imaging (comparing standard and experimental high resolution diffusion-weighted imaging [DWI] MRI with 18F-Fluciclovine)
  Other Names: Axumin; prostate-cancer-specific radiotracer

SUMMARY:
This prospective trial aims to determine if enhanced prostate imaging using two novel imaging technologies (high resolution DWI and 18F-fluciclovine PET-MRI) will detect prostate cancers not seen on standard multiparametric prostate MRI in patients considered candidates for focal HIFU.

DETAILED DESCRIPTION:
This is a prospective trial to evaluate the effectiveness of 18F-fluciclovine PET-hrMRI versus standard mpMRI at identifying prostate cancer targets for HIFU therapy.

Participants with clinically localized, unilateral high grade prostate cancer (Gleason score 7-10 prostate cancer localized to one lobe on prior biopsies) OR at high risk for having unrecognized high grade prostate cancer (overall Gleason score 6 with > half of systematic biopsy cores positive and > 50% of core involvement in at least one core), interested in HIFU would receive both a standard mpMRI and 18F-fluciclovine PET-hrMRI.

Participants would then undergo a mapping biopsy using a standard sextant template plus MRI/US-fusion targeted biopsy of any lesion suspicious lesion on mpMRI or PET-hrMRI.

ELIGIBILITY:
Inclusion Criteria:

* Prostate biopsy consisting of ≥ 10 tissue cores sampled
* PSA </=20 ng/mL
* cT1-cT2c
* Either overall gleason score >/= 7 with Gleason grade 4 or 5 component localized to one lobe (i.e. right or left) OR overall Gleason score 6 with >/= half of systematic biopsy cores positive and >/= 50% of core involvement in at least one core
* Patient considering focal HIFU therapy

Exclusion Criteria:

* Previous local therapy for prostate cancer
* Inability to receive PET tracer
* Inability to receive MRI
* Suggestion of extracapsular extension or seminal vesicle invasion on imaging
* Estimated creatinine clearance <45 mL/min (Cockcroft-Gault equation)
* Any other condition which, in the investigator's option, may make the patient a poor candidate for participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Daskivich, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Opened to accrual on 12/07/2017 with first subject enrolled on study 12/18/2017. A total of 21 patients consented, one withdrew consent prior to intervention and was replaced, 13 were evaluable for primary outcome measure, however 11 subjects of the total target accrual of 20 subjects completed study with the last subject off treatment/off study as of 1/8/2020.
Groups:
- 18F-Fluciclovine: 10mCi +/-20% 18F-fluciclovine injection
  18F-Fluciclovine: Imaging (comparing standard and experimental high resolution diffusion-weighted imaging [DWI] MRI with 18F-Fluciclovine)
  Prior to HIFU therapy, all subjects undergo mapping MRI using both standard mpMRI and experimental diffusion-weighted imaging (DWI) PET-hrMRI with 18F-Fluciclovine. PET scans involve injection of the radioisotope or tracer, where all subjects will receive 10mCi +/-20% 18F-fluciclovine injection, diluted up to 10mL injected via the IV, as an IV bolus injection followed by 10mL flush with normal saline solution.
Period: Overall Study
Arm/Group | 18F-Fluciclovine
Started | 21
Completed | 11 (13 evaluable for primary outcome, but 11 total completed study.)
Not Completed | 10
Not completed — Withdrawal by Subject | 3
Not completed — Ineligible (incomplete post-HIFU) | 7

BASELINE CHARACTERISTICS:
Arm/Group | 18F-Fluciclovine
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 70 [51 to 77]
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Biopsy-proven Cancers (Gleason 6+) That Standard Imaging (mpMRI) Would Have Missed Compared With High Resolution Diffusion-weighted Imaging (DWI) PET-hrMRI on Mapping MRI.
Description: A Gleason score of 6 is low grade, 7 is intermediate grade, and a score of 8 to 10 is high grade cancer. The Prostate Imaging Reporting and Data System (PI-RADS) is used to report how likely it is that a suspicious area is a clinically significant cancer. PI-RADS scores range from 1 (most likely not cancer) to 5 (very suspicious). Difference between sensitivities to identify prostate lesions. This is analyzed by the number of biopsy-proven cancerous zones (Gleason 6+) that mpMRI missed compared to PET or hrMRI (PIRADS) compared as follows:
  mpMRI vs hrMRI and PET (PIRADS 3-5 & Gleason 7+) mpMRI vs hrMRI or PET (PIRADS 3-5 & Gleason 7+)
  mpMRI vs hrMRI and PET (PIRADS 4-5 & Gleason 7+) mpMRI vs hrMRI or PET (PIRADS 4-5 & Gleason 7+)
  mpMRI vs hrMRI and PET (PIRADS 3-5 & Gleason 6+) mpMRI vs hrMRI or PET (PIRADS 3-5 & Gleason 6+)
  mpMRI vs hrMRI and PET (PIRADS 4-5 & Gleason 6+) mpMRI vs hrMRI or PET (PIRADS 4-5 & Gleason 6+)
Time Frame: At time of post-imaging biopsy
Measure: Number; unit: Total biopsy-proven cancers (Gleason 6+)
Units Other Than Participants: Total biopsy-proven cancers (Gleason 6+)
Arm/Group | 18F-Fluciclovine
Number analyzed (Participants) | 13
Number analyzed (Total biopsy-proven cancers (Gleason 6+)) | 32
Total biopsy-proven cancers (Gleason 6+)
  Number of biopsy-proven cancers (Gleason 6+) that mpMRI missed compared to PET or hrMRI (PIRADS 3-5) | 5
  Number of biopsy-proven cancers (Gleason 6+) that mpMRI missed compared to PET & hrMRI (PIRADS 3-5) | 1
  Number of biopsy-proven cancers (Gleason 6+) that mpMRI missed compared to PET or hrMRI (PIRADS 4-5) | 4
  Number of biopsy-proven cancers (Gleason 6+) that mpMRI missed compared to PET & hrMRI (PIRADS 4-5) | 1
Statistical Analysis 1: Comparison: 18F-Fluciclovine; mpMRI vs hrMRI and PET (PIRADS 3-5 & Gleason 6+); Test type: Superiority; p = 0.056, Durkalski's Chi-square test — mpMRI vs hrMRI and PET (PIRADS 3-5 & Gleason 6+); Sensitivity = 0.25, 95% CI 2-sided [0.19 to 0.46] — We did not present standard deviation as the variability is already incorporated in the provided confidence interval
Statistical Analysis 2: Comparison: 18F-Fluciclovine; mpMRI vs hrMRI or PET (PIRADS 3-5 & Gleason 6+); Test type: Superiority; p = 0.56, Durkalski's Chi-square test — mpMRI vs hrMRI or PET (PIRADS 3-5 & Gleason 6+); Sensitivity = 0.56, 95% CI 2-sided [0.44 to 0.78] — We did not present standard deviation as the variability is already incorporated in the provided confidence interval
Statistical Analysis 3: Comparison: 18F-Fluciclovine; mpMRI vs hrMRI and PET (PIRADS 4-5 & Gleason 6+); Test type: Superiority; p = 0.060, Durkalski's Chi-square test — mpMRI vs hrMRI and PET (PIRADS 4-5 & Gleason 6+); Sensitivity = 0.22, 95% CI 2-sided [0.17 to 0.47] — We did not present standard deviation as the variability is already incorporated in the provided confidence interval
Statistical Analysis 4: Comparison: 18F-Fluciclovine; mpMRI vs hrMRI or PET (PIRADS 4-5 & Gleason 6+); Test type: Superiority; p = 0.083, Durkalski's Chi-square test — mpMRI vs hrMRI or PET (PIRADS 4-5 & Gleason 6+); Sensitivity = 0.50, 95% CI 2-sided [0.39 to 0.74] — We did not present standard deviation as the variability is already incorporated in the provided confidence interval

2. Primary Outcome: Number of Biopsy-proven Cancers (Gleason 7+) That Standard Imaging (mpMRI) Would Have Missed Compared With High Resolution Diffusion-weighted Imaging (DWI) PET-hrMRI on Mapping MRI.
Description: A Gleason score of 6 is low grade, 7 is intermediate grade, and a score of 8 to 10 is high grade cancer. The Prostate Imaging Reporting and Data System (PI-RADS) is used to report how likely it is that a suspicious area is a clinically significant cancer. PI-RADS scores range from 1 (most likely not cancer) to 5 (very suspicious). Difference between sensitivities to identify prostate lesions. This is analyzed by the number of biopsy-proven cancerous zones (Gleason 7+) that mpMRI missed compared to PET or hrMRI (PIRADS) compared as follows:
  mpMRI vs hrMRI and PET (PIRADS 3-5 & Gleason 7+) mpMRI vs hrMRI or PET (PIRADS 3-5 & Gleason 7+)
  mpMRI vs hrMRI and PET (PIRADS 4-5 & Gleason 7+) mpMRI vs hrMRI or PET (PIRADS 4-5 & Gleason 7+)
  mpMRI vs hrMRI and PET (PIRADS 3-5 & Gleason 6+) mpMRI vs hrMRI or PET (PIRADS 3-5 & Gleason 6+)
  mpMRI vs hrMRI and PET (PIRADS 4-5 & Gleason 6+) mpMRI vs hrMRI or PET (PIRADS 4-5 & Gleason 6+)
Time Frame: At time of post-imaging biopsy
Measure: Number; unit: Total biopsy-proven cancers (Gleason 7+)
Units Other Than Participants: Total biopsy-proven cancers (Gleason 7+)
Arm/Group | 18F-Fluciclovine
Number analyzed (Participants) | 13
Number analyzed (Total biopsy-proven cancers (Gleason 7+)) | 20
Total biopsy-proven cancers (Gleason 7+)
  Number of biopsy-proven cancers (Gleason 7+) that mpMRI missed compared to PET or hrMRI (PIRADS 3-5) | 1
  Number of biopsy-proven cancers (Gleason 7+) that mpMRI missed compared to PET & hrMRI (PIRADS 3-5) | 1
  Number of biopsy-proven cancers (Gleason 7+) that mpMRI missed compared to PET or hrMRI (PIRADS 4-5) | 1
  Number of biopsy-proven cancers (Gleason 7+) that mpMRI missed compared to PET & hrMRI (PIRADS 4-5) | 1
Statistical Analysis 1: Comparison: 18F-Fluciclovine; mpMRI vs hrMRI and PET (PIRADS 3-5 & Gleason 7+); Test type: Superiority; p = 0.096, Durkalski's Chi-square test — mpMRI vs hrMRI and PET (PIRADS 3-5 & Gleason 7+); Sensitivity = 0.35, 95% CI 2-sided [0.26 to 0.65] — We did not present standard deviation as the variability is already incorporated in the provided confidence interval
Statistical Analysis 2: Comparison: 18F-Fluciclovine; mpMRI vs hrMRI or PET (PIRADS 3-5 & Gleason 7+); Test type: Superiority; p = 0.317, Durkalski's Chi-square test — mpMRI vs hrMRI or PET (PIRADS 3-5 & Gleason 7+); Sensitivity = 0.60, 95% CI 2-sided [0.46 to 0.90] — We did not present standard deviation as the variability is already incorporated in the provided confidence interval
Statistical Analysis 3: Comparison: 18F-Fluciclovine; mpMRI vs hrMRI and PET (PIRADS 4-5 & Gleason 7+); Test type: Superiority; p = 0.063, Durkalski's Chi-square test — mpMRI vs hrMRI and PET (PIRADS 4-5 & Gleason 7+); Sensitivity = 0.30, 95% CI 2-sided [0.23 to 0.66] — We did not present standard deviation as the variability is already incorporated in the provided confidence interval
Statistical Analysis 4: Comparison: 18F-Fluciclovine; mpMRI vs hrMRI or PET (PIRADS 4-5 & Gleason 7+); Test type: Superiority; p = 0.317, Durkalski's Chi-square test — mpMRI vs hrMRI or PET (PIRADS 4-5 & Gleason 7+); Sensitivity = 0.60, 95% CI 2-sided [0.46 to 0.90] — We did not present standard deviation as the variability is already incorporated in the provided confidence interval

3. Secondary Outcome: Negative Biopsy Rate (Number of Participants With Negative Biopsy)
Description: A Gleason score of 6 is low grade, 7 is intermediate grade, and a score of 8 to 10 is high grade cancer. The Prostate Imaging Reporting and Data System (PI-RADS) is used to report how likely it is that a suspicious area is a clinically significant cancer. PI-RADS scores range from 1 (most likely not cancer) to 5 (very suspicious). Following the tumor mapping study, patients with high grade disease (i.e. Gleason grade 4 or 5) in one lobe undergo hemigland or focal HIFU of that lobe. Patients would then undergo repeat prostate biopsy to assess the negative biopsy rate in the treated region.
Time Frame: 6 months following standard HIFU therapy
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-Fluciclovine
Number analyzed (Participants) | 13
Participants | 11

4. Secondary Outcome: Rate of High Grade Cancer (Number of Patients With High Grade Cancer)
Description: A Gleason score of 6 is low grade, 7 is intermediate grade, and a score of 8 to 10 is high grade cancer. The Prostate Imaging Reporting and Data System (PI-RADS) is used to report how likely it is that a suspicious area is a clinically significant cancer. PI-RADS scores range from 1 (most likely not cancer) to 5 (very suspicious). Following the tumor mapping study, patients with high grade disease (i.e. Gleason grade 4 or 5) in one lobe undergo hemigland or focal HIFU of that lobe. Patients would then undergo repeat prostate biopsy to assess the absence of Gleason grade 4 or 5 in the untreated region.
Time Frame: 6 months following standard HIFU therapy
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-Fluciclovine
Number analyzed (Participants) | 11
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 6 months following standard HIFU therapy.
Arm/Group | 18F-Fluciclovine
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-Fluciclovine (N=13)
Sepsis (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT03263780/Prot_SAP_001.pdf